CLINICAL TRIAL: NCT07077317
Title: Examining the Effects of the Stop-Bang Scoring Model, Anthropometric Measurements, and Head Dimensions on Difficult Airway Prediction
Brief Title: Examining the Effects of Anthropometric Measurements on Difficult Airway Prediction
Status: Completed | Type: Observational
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Suleyman Camgoz, Asistant Professor, Kutahya Health Sciences University
Other Study IDs: E-41997688-050.99-177377
Record Dates: First submitted 2025-07-11; First posted 2025-07-22 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Difficult Airway; Difficult Airway Intubation; Airway Management
Keywords: mask ventilation; intubation; Cormack-Lehane; Airway Assessment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Airway Assessment Using Standard Clinical Tools — Preoperative airway evaluation using routine physical measurements (e.g., Mallampati score, neck circumference, STOP-Bang questionnaire), and intraoperative/postoperative observation of airway-related parameters.

SUMMARY:
Airway-related complications are among the leading causes of anesthesia-associated morbidity and mortality. Therefore, the ability to predict difficult mask ventilation, laryngoscopy, and intubation before induction is essential to ensure proper preparation in patients at risk and avoid unnecessary airway manipulations in low-risk individuals. While numerous studies have focused on predicting difficult intubation, most have limited sample sizes and do not consider postoperative critical respiratory events.

In this prospective observational clinical study, we aim to investigate the relationship between commonly used preoperative airway assessment tools-including anthropometric measurements, Mallampati score, and the STOP-Bang questionnaire for obstructive sleep apnea-and the incidence of difficult mask ventilation, difficult laryngoscopy (Cormack-Lehane grading), difficult intubation, and critical respiratory events in the postoperative period.

The study will include adult patients (≥18 years) classified as ASA I-IV undergoing surgery under general anesthesia with endotracheal intubation. Data will be collected preoperatively, intraoperatively, and in the post-anesthesia care unit (PACU) by experienced anesthesia personnel. Postoperative critical respiratory events are defined as unexpected hypoxemia, hypoventilation, reintubation, or interventions required for upper/lower airway obstruction.

DETAILED DESCRIPTION:
Difficult airway management remains one of the most significant challenges in clinical anesthesia, often leading to severe complications such as hypoxemia, aspiration, and even cardiac arrest. Despite various clinical predictors, no single assessment method reliably identifies all patients at risk. This prospective, observational study aims to comprehensively evaluate the association between preoperative airway assessment parameters and both intraoperative airway difficulty and postoperative critical respiratory events.

The preoperative assessment will include demographic characteristics, comorbidities, ASA classification, Mallampati score, and detailed anthropometric airway measurements (neck circumference, thyromental distance, sternomental distance, interincisor gap, head dimensions, presence of beard/dentition, and neck mobility). Additionally, the STOP-Bang questionnaire will be administered to assess the risk of obstructive sleep apnea (OSA).

During induction and airway management, mask ventilation difficulty will be graded, Cormack-Lehane score during laryngoscopy will be recorded, and intubation will be evaluated in terms of the number of attempts and need for adjunctive devices (stylet, bougie, fiberoptic bronchoscope, videolaryngoscope, etc.).

In the postoperative phase, patients will be monitored for critical respiratory events including unexpected hypoxemia (SpO₂ <90%), hypoventilation (RR <8/min or PaCO₂ >50 mmHg), reintubation, and any interventions (e.g., airway support, bronchodilators, cold mist, etc.) required for upper or lower airway obstruction.

The outcomes of this study may help refine preoperative screening protocols and contribute to the development of risk-based airway management strategies aimed at improving patient safety.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years,
* ASA Physical Status I, II, III or IV,
* Undergoing elective surgery under general anesthesia with endotracheal intubation,
* Written informed consent provided

Exclusion Criteria:

* History of head and neck surgery or trauma causing anatomical deformity,
* Known congenital or acquired airway abnormality,
* Cervical spine surgery or instability,
* Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing elective surgical procedures requiring endotracheal intubation under general anesthesia at a tertiary hospital.
Sampling Method: Non-Probability Sample
Enrollment: 1044 (Actual)
Dates: Start 2025-08-13 (Actual); Primary Completion 2025-10-30 (Actual); Study Completion 2025-11-11 (Actual)

PRIMARY OUTCOMES:
Incidence of Difficult Mask Ventilation | Intraoperative (during anesthesia induction)
  Evaluation of mask ventilation using a standard difficulty grading scale.
  1. Mask Ventilation Successful
  2. Mask Ventilation Requires Oral Airway
  3. Mask Ventilation Requires Oral Airway And Assistant (Two Hands)
  4. Mask Ventilation Failure
Incidence of Difficult Laryngoscopy | Intraoperative (during laryngoscopy)
  Cormack-Lehane grade III-IV views considered difficult laryngoscopy.
Incidence of Difficult Intubation | Intraoperative (during intubation)
  Defined as more than two attempts, or the requirement of adjuncts such as bougie, videolaryngoscope, or fiberoptic bronchoscope.
Occurrence of Postoperative Critical Respiratory Events | Within the first 2 hours postoperatively (in PACU)
  Events include unexpected hypoxemia (SpO₂ < 90%), hypoventilation (RR < 8/min or PaCO₂ > 50 mmHg), reintubation, and active interventions for airway obstruction.

SECONDARY OUTCOMES:
Correlation Between STOP-Bang Score and Difficult Airway Incidence | Preoperative through intraoperative period
  Evaluate predictive value of high STOP-Bang scores (≥3) for difficult mask ventilation, laryngoscopy, and intubation.
Correlation Between Anthropometric Measurements and Critical Respiratory Events | Preoperative to postoperative period
  Investigate associations between variables such as neck circumference, interincisor gap, or sternomental distance with postoperative respiratory complications.
Correlation Between Anthropometric Measurements and Difficult Airway Management | Preoperative to intraoperative (induction period of anesthesia)
  Investigate associations between variables such as neck circumference, interincisor gap, or sternomental distance, head dimensions, with difficult mask ventilation or difficult intubation.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology, KUTAHYA CITY HOSPITAL, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No